CLINICAL TRIAL: NCT05243069
Title: Head and Neck Cancer Patient Symptom and Oncologic Outcomes as a Function of Head and Neck Volume Changes
Brief Title: Head and Neck Cancer Patient Symptom and Oncologic Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Roman Skoracki, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OSU-20210; NCI-2020-08318 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-02-24; First posted 2022-02-16 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: Lymphedema of the Head and Neck
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening (3D scan) (Experimental): Patients undergo 3D scanning of lower head and neck region over 90-120 seconds before surgery and then every 3 months for up to 1 year after surgery.
  Interventions: Procedure: Imaging Technique

INTERVENTIONS:
Procedure: Imaging Technique — Undergo 3D scanning
  Other Names: Diagnostic Imaging Technique; Imaging; imaging procedure; Imaging Procedures; Imaging, Not Otherwise Specified; Medical Imaging

SUMMARY:
This trial investigates a new approach using a mobile three-dimensional (3D) scanning application for volumetric measurement of the head and neck region in patients with head and neck lymphedema. Lymphedema is the buildup of extra lymph fluid in tissues that causes swelling. Accurate volumetric measurements of swelling are crucial to the diagnosis of lymphedema and to monitoring response to therapy and disease progression over time. A mobile 3D surface scanning application may help doctors measure and analyze swelling in patients with head and neck lymphedema.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a specialized and mobile 3D surface scanning application to assess and monitor head and neck lymphedema.

II. To confirm optimal positioning when volumetrically assessing head and neck lymphedema using 3D technologies as consistent with standard plastic surgery departmental protocol.

III. To quantify and serially track changes in head and neck lymphedema in patients with pathologies and correlate these changes with overall patient well-being and disease progression.

OUTLINE:

Patients undergo 3D scanning of lower head and neck region over 90-120 seconds before surgery and then every 3 months for up to 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologies leading to head and neck lymphedema
* Individuals with minimal or no facial hair
* Patients of sound mentation, who are able to execute informed decision-making

Exclusion Criteria:

* Any health conditions or history of non-compliance that affect the study will preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Volume of interest between the cutting planes | Up to 24 weeks
  Will examine the volume of interest between the cutting planes that are determined by the anatomical landmarks around the eyebrows, ears and jaw that are manually identified from the three-dimensional (3D) surface scans. The volume of interest will be calculated for each 3D scan by a computer algorithm developed by Knockout Concepts. Test-rest reliability will be assessed by concordance correlation coefficients with 95% confidence interval by comparing two sets of volume of interest between repeated scans at each encounter. In addition, Bland-Altman plots with 95% Limits of Agreement will be reported for the bias between the two scoring systems.
Average values of the two repeated scans | Up to 24 weeks
  Average values of the two repeated scans at each encounter will be plotted over the five clinical visits to graphically explore the trajectory of the change in the primary outcome.
Patient wellbeing/disease progression | Up to 24 weeks
  Correlation between head and neck lymphedema and patient wellbeing/disease progression will be done by using linear regression, Pearson's correlation coefficient or spearman's correlation coefficient, depending on the distribution of the data.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Skoracki, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu